CLINICAL TRIAL: NCT06102564
Title: GST-moms: Effects of Group-schematherapy on Mother-child Attachment
Brief Title: GST-moms: Effects of Group-schematherapy on Mother-child Attachment Relations
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Maastricht University (Other)
Collaborators: Psychologiepraktijk Esra (Unknown)
Responsible Party: Principal Investigator, Jeffrey Roelofs, Principal Investigator/Clinical professor (PhD), Maastricht University
Other Study IDs: ERCPN 264_29_02_2023
Record Dates: First submitted 2023-04-13; First posted 2023-10-26 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Cluster C Personality Disorder (Diagnosis); Mother-Child Relations
Keywords: Group Schematherapy; Mother-child attachment; Effectiviness
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Group schematherapy — Brief group schematherapy for mothers with young children (age 0-5) focused on attachment relations between mother and child

SUMMARY:
The birth of a baby can be a stressful period. Dysfunctional schemas of the 'new' parent can be triggered making it more difficult to discern what the baby needs are. In schema therapy terms, mentalizing capacity is best described as the "healthy adult mode". A parent who responds to her baby from a healthy adult mode provides the baby a safe environment for self-development. However, interpreting the baby's signals can be a constant challenge for some parents. This can trigger early attachment relationships and schemas. At such times, the parent may become overwhelmed by their own emotions and respond less adequate to the child's needs. Distorted parental reflective functioning is associated both with insecure attachment and poor affect regulation in the parent and with various psychological disorders in the child. Treatments aimed at improving parental reflectiveness seem to have a positive impact on the quality of the attachment between parents and their baby.

The objective of this study is to measure the effects of the group-schematherapy for mothers with young children (GST moms) on mother-child attachment relations. The aim is to help moms regulate their own emotions, by understanding their own modes and schema's. In doing so will help them feel more confident to mentalize about their child and to adequately respond to their needs and emotionally bond with their baby. The researchers anticipate it will improve the quality of attachment between mother and child. Many studies have been done on the effectiveness of group schematherapy however there are no studies specifically for schematherapy for parents, in this case mothers. GST moms can be an early intervention aimed at prevention of psychological problems with the child.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients for the group schematherapy are mothers with young children (0-5 years), with a cluster C personality disorder.

Exclusion Criteria:

* Acute Suicidal or chronic suicidality
* Psychotic disorder
* Autistic spectrum disorder
* Bipolar disorder
* Developmental disorders
* Any other AS-I disorder that requires treatment first (severe depression, alcohol and/or drugs abuse)
* Cluster A or B personality disorders (traits of cluster B in combination with Cluster C personality disorder is included)
* Neuropsychological damage
* General problems for group therapy (auditory impairment, severe physical disability, insufficant Dutch comprehension, IQ < 80)
* Self-mutilation

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Mothers with young children (0-5 years) with Cluster C personality disorder or mixed/other personality disorder (cluster C and cluster B traits) who encounter problems in the mother-child interaction. They may have depressive and/or anxiety symptoms aswell.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The Maternal Postnatal attachment Scale (MPAS, 2015) | Inclusion (week 1), start therapy (variable; at least 20 weeks after inclusion), evaluation (week 10), end of group therapy (week 20), follow-up (3 months completion = week 20)
  A 19 item self-report questionnaire that is used to assess mother-to-infant attachment (theemotional bond or affection experienced by the parent towards the infant)
The Parental Reflective Functioning Questionnaire (PRFQ, 2009) | Inclusion (week 1), start therapy (variable; at least 20 weeks after inclusion), evaluation (week 10), end of group therapy (week 20), follow-up (3 months completion = week 20)
  A self-report instrument of reflective functioning.

SECONDARY OUTCOMES:
The Young Schema Questionnaire YSQ-S3 (YSQ-S3; Young, 1994). | Inclusion (week 1), start therapy (variable; at least 20 weeks after inclusion), evaluation (week 10), end of group therapy (week 20), follow-up (3 months completion = week 20)
  De Young Schema Questionnaire is a self-report instrument to assess 18 dysfunctional schemas and consists of 90 items
The Schema Mode Inventory (SMI, Lobbestael, 2017) | Inclusion (week 1), start therapy (variable; at least 20 weeks after inclusion), evaluation (week 10), end of group therapy (week 20), follow-up (3 months completion = week 20)
  To asses schema modes (118 items)
Brief Sympthom Inventory (BSI, Derogatis, 1975, de Beurs, 2006) | Inclusion (week 1), start therapy (variable; at least 20 weeks after inclusion), evaluation (week 10), end of group therapy (week 20), follow-up (3 months completion = week 20)
  A self-report questionnaire to evaluate a broad range of psychological problems and symptoms of psychopathology.
The Beck Depression Inventory (BDI; Beck et al., 1996) | Inclusion (week 1), start therapy (variable; at least 20 weeks after inclusion), evaluation (week 10), end of group therapy (week 20), follow-up (3 months completion = week 20)
  A self-report questionnaire of depressive symptoms.

OTHER OUTCOMES:
The Working Model of the child interview (WMCI; Zeanah, Benoit & Barton, 1996) | Inclusion Week 1
  The WMCI is a semistructured interview to asses the internal representations of their child and relationship with the child.
The Childhood Trauma Questionnaire (CTQ; Bernstein, 1994) | Inclusion Week 1
  A self report measure to identify diffent types of childhood trauma and abuse.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Roelofs, PhD, Principal Investigator — Maastricht University